CLINICAL TRIAL: NCT06403553
Title: The Dynamic Change of Fecal Calprotectin From Day 1 to Day 3 Was Associated With Sepsis-associated Liver Dysfunction
Brief Title: FC Change From Day 1 to Day 3 Associated With SALD
Acronym: 2024-04-22
Status: Completed | Type: Observational
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: 2024-04-22
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-01

CONDITIONS: Liver Dysfunction
Keywords: Sepsis-associated Liver Dysfunction
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-SALD group: patients does not fulfill any of the following conditions during ICU stay:
  1. Serum aminotransaminase levels > 800 IU/L, including alanine aminotransferase and aspartate aminotransferase;
  2. Total bilirubin > 2 mg/dL.
  Interventions: Diagnostic Test: Fecal Calprotectin
- SALD group: when patients meet either of the following two criteria under sepsis condition during ICU stay:
  1. Serum aminotransaminase levels > 800 IU/L, including alanine aminotransferase and aspartate aminotransferase;
  2. Total bilirubin > 2 mg/dL.
  Interventions: Diagnostic Test: Fecal Calprotectin

INTERVENTIONS:
Diagnostic Test: Fecal Calprotectin — Fecal Calprotectin measurement on days 1and 3

SUMMARY:
As defined by sepsis 3.0, sepsis is a clinical syndrome caused by disordered host response to serious infection，leading to multiple organ dysfunction1. Sepsis-associated liver dysfunction (SALD) is one of the most frequently complication in sepsis, possessing high morbidity and mortality2.

A close relationship exists between the gut and the liver, and their bidirectional interaction was commonly known as the 'gut-liver' axis3. Systemic inflammation and hypoperfusion play a crucial role in the pathophysiological processes of acute gastrointestinal injury (AGI) in sepsis4. The translocation of bacteria and toxins due to gut barrier injury during AGI can promote the entry of bacteria and their products into the liver through the portal circulation and lymphatic system, leading to the occurrence of SALD. Our previous study found that septic patients with abdominal infections and SALD suffered a higher incidence of AGI when compared with patients without SALD5.

Faecal calprotectin (FC) is a convenient, non-invasive biomarker that has a good correlation with gut inflammation6. The FC concentration is proportional to neutrophil migration to the gut and correlates well with fecal leukocyte excretion7. Study found that FC concentrations were significantly higher in septic patients complicated with AGI than those without, and it can be used as an early indicator for the diagnosis of AGI8. However, the relationship between FC concentration and SALD in septic patient is unclear. We conducted a prospective study to explore the potential association between FC concentration and SALD in septic patients. The dynamic changes in the FC concentration from day 1 to 3 after enrollment were also investigated.

DETAILED DESCRIPTION:
Study participants

This was a single-center prospective observational study enrolling consecutive adult patients with sepsis (≥18 years) admitted to Nanjing Drum Tower Hospital between January 2023 to March 2024. The study protocol was approved by the Medical Ethics Committee of local institution (number: 2023-396-03). All patients or their immediate family members provided the informed consent and all study procedures were in line with the Declaration of Helsinki. Exclusion criteria were:

1. had diseases originating in the gastrointestinal tract, such as gastrointestinal malignancies and inflammatory bowel disease (IBD);
2. complicated by severe chronic liver diseases, such as decompensated cirrhosis and advanced liver cancer;
3. hospitalization for primary hepatobiliary disease, such as trauma, hepatitis and hepatic abscess;
4. already diagnosed SALD at enrollment;
5. were discharged or died within 72 hours after enrollment;
6. were pregnant.

All eligible patients were treated according to the sepsis 3.0 guidelines, including: control the source of infection, used antibiotic early and other supportive therapies to maintain organ function. Patients were divided into non-SALD and SALD groups according to SALD whether or not diagnosed during intensive care units (ICU) stay. Eligible patients also be excluded if the following occurs during the study period:

1. deviation from the study protocol for any reason;
2. have other causes of liver injury, such as drugs and poisons;
3. diagnosis of SALD within 72 hours after enrollment;
4. patients or their relatives decided to withdraw from the study.

Data collection and outcomes The primary study outcome was the FC concentration (<50.00 μg/g), which reflect the severity of gut inflammation. Fecal samples were collected from patients on days 1 and 3 after inclusion using sterile tubes and stored at 4°C, and FC was measured within 48 hours of collection using commercial ELISA (KAPEPKT849, Beijing North Institute of Biotechnology Co.,Ltd., Beijing, China) following the manufacturer's instruction. The following information were collected within the first 24 hours of enrollment, including: demographic characteristics, including age, gender and comorbidity; the sources of infection; disease severity scores, including Acute Physiology and Chronic Health Evaluation (APACHE) II score and Sequential Organ Failure Assessment (SOFA) score; complications, including respiratory failure, septic shock, acute kidney injury (AKI), and AGI; inflammatory factors, including interleukin (IL)-1β,IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-17, interferon (IFN)-α，IFN-γand tumor necrosis factor (TNF); other indicators, including human leukocyte antigen (HLA)-DR, albumin, platelet and D-dimer were also recorded. The following indicators were collected on days 1 and 3 after enrollment: white blood cell (WBC) count, neutrophil count, lymphocyte count, C-reactive protein, procalcitonin and IL-6. Prognostic indicators included ICU length of stay (LOS) and ICU mortality were also recorded.

Definitions

Sepsis and septic shock were diagnosed based on criteria established by the Sepsis 3.0 guidelines1. SALD was diagnosed when patients meet either of the following two criteria under sepsis condition9:

1. Serum aminotransaminase levels > 800 IU/L, including alanine aminotransferase and aspartate aminotransferase;
2. Total bilirubin > 2 mg/dL. AKI was diagnosed in accordance with the Kidney Disease Improving Global Outcomes clinical practice guidelines10. The diagnosis of AGI was based on the ESICM recommendations in 201211. The term 'FC1' was used to represent the FC concentration on day 1 and 'FC3' on day 3. The term 'ΔFC' was used to represent the concentration of the FC3 minus the concentration of the FC1.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with sepsis

Exclusion Criteria:

* had diseases originating in the gastrointestinal tract, such as gastrointestinal malignancies and inflammatory bowel disease (IBD);
* complicated by severe chronic liver diseases, such as decompensated cirrhosis and advanced liver cancer;
* hospitalization for primary hepatobiliary disease, such as trauma, hepatitis and hepatic abscess;
* already diagnosed SALD at enrollment;
* were discharged or died within 72 hours after enrollment;
* were pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients were treated according to the sepsis 3.0 guidelines, including: control the source of infection, used antibiotic early and other supportive therapies to maintain organ function. Patients were divided into non-SALD and SALD groups according to SALD whether or not diagnosed during intensive care units (ICU) stay. Eligible patients also be excluded if the following occurs during the study period:
  1. deviation from the study protocol for any reason;
  2. have other causes of liver injury, such as drugs and poisons;
  3. diagnosis of SALD within 72 hours after enrollment;
  4. patients or their relatives decided to withdraw from the study.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of SALD | 30 days after ICU admission
  whether SALD occurs

SECONDARY OUTCOMES:
mortality | 30 days after ICU admission
  death or not

CONTACTS AND LOCATIONS:
Locations (1):
- Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
There is another study currently sharing relevant information

REFERENCES:
- [Background] Zhang B, Chen X, He C, Su T, Cao K, Li X, Duan J, Chen M, Zhu Z, Yu W. Acute gastrointestinal injury and altered gut microbiota are related to sepsis-induced cholestasis in patients with intra-abdominal infection: a retrospective and prospective observational study. Front Med (Lausanne). 2023 Jul 27;10:1144786. doi: 10.3389/fmed.2023.1144786. eCollection 2023. PMID 37575984
- [Result] Li J, Ren Y, Gao C, Zhang K, Zheng F, Kang J. Evaluation of Fecal Calprotectin, D-Lactic Acid and Bedside Gastrointestinal Ultrasound Image Data for the Prediction of Acute Gastrointestinal Injury in Sepsis Patients. Front Med Technol. 2021 Nov 1;3:733940. doi: 10.3389/fmedt.2021.733940. eCollection 2021. PMID 35047957